CLINICAL TRIAL: NCT02821364
Title: Philadelphia Immediate Transport in Penetrating Trauma Trial
Acronym: PIPT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not feasible due to logistical elements
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 22749
Record Dates: First submitted 2016-04-13; First posted 2016-07-01 (Estimated); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Hemorrhagic Shock; Peritonitis
MeSH Terms: conditions — Shock, Hemorrhagic; Peritonitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Life Support (Other): ALS providers are trained and able to perform certain procedures such as intubation with endotracheal tubes and placement of intravenous catheters. Endotracheal intubation is often performed by pre-hospital providers in critically ill trauma patients because it is believed that it allows for protection of the airway and better delivery of oxygen. However, most studies actually show that intubation does not provide a survival advantage to this patient population and actually could result in worse outcomes. Intravenous catheter placement and administration of intravenous fluids is also routinely performed however, studies have shown that it is also not helpful.
  Interventions: Other: Advanced Life Support
- Basic Life Support (No Intervention): Subjects randomized to the study group will receive basic life support (BLS) level care. This means that pre-hospital procedures such as endotracheal intubation and intravenous fluid administration will not be carried out. However, passive oxygen and needle thoracostomy, if required for tension pneumothorax, will be permitted if medically necessary.

INTERVENTIONS:
Other: Advanced Life Support — IV FLUIDS, INTUBATION
  Arms: Advanced Life Support

SUMMARY:
PIPT Trial (Philadelphia Immediate Transport in Penetrating Trauma Trial) A prospective randomized clinical trial comparing pre-hospital procedures to immediate transportation in patients with penetrating injury and shock.

DETAILED DESCRIPTION:
The establishment of Advanced Life Support by emergency medical services (EMS) has led to an increasing number of procedures being carried out in the field. These procedures, such as intravenous (IV) fluid administration and endotracheal intubation can be beneficial in rural settings where transportation to definitive care is prolonged. In addition, it can provide benefit to patients with traumatic brain injury. However, data on field procedures carried out in penetrating trauma patients in urban locations is less convincing and actually shows that these procedures result in worse morbidity and mortality, where penetrating injury is defined as resulting from gunshot, shotgun or stab wounds. In fact, studies have shown that pre-hospital intubation clearly does not confer a survival advantage to penetrating trauma patients in urban locations. Yet pre-hospital procedures continue to be performed in urban Philadelphia on a regular basis. In a recently published study at Temple University Hospital from 2006-2010, of the 1,615 gunshot and stab wound victims that were highest level trauma activations, 152 (9.8%) were intubated in the field. In another study carried out at Temple University Hospital looking at the most critically ill penetrating trauma patients that required emergency room thoracotomy, 71.8% of patients transported by EMS were intubated and 67.0% received IV fluids. This demonstrates that these procedures are being carried out with regularity in severely injured penetrating trauma patients.

Patient recruitment and randomization will occur at the time that the distress call is received by the EMS dispatcher and an ALS crew is dispatched. The dispatcher will assign the patient to advanced life support current practice or immediate transport with basic life support current practice based on even or odd dispatch number. All participating paramedics will be given face to face training in the conduct of the trial, and provided with resources for online refreshers and reminders. Compliance with enrollment procedures will be monitored through redundant mechanisms including notification at hospital arrival, cross referenced to monthly monitoring of EMS reports.

Subjects randomized to the study group will receive basic life support (BLS) level care. This means that pre-hospital procedures such as endotracheal intubation and intravenous fluid administration will not be carried out. However, passive oxygen and needle thoracostomy, if required for tension pneumothorax, will be permitted if medically necessary. For patients in the control group, ALS responders will perform advanced life support current practice, including intravenous fluid administration and endotracheal intubation as deemed appropriate.

ELIGIBILITY:
Inclusion Criteria:

The investigators will include all penetrating trauma patients with shock over the age of 18.

1. Penetrating injury (required)
2. Combined torso and distal extremity injury
3. Combined penetrating and blunt injury
4. Heart rate greater than 100, systolic blood pressure less than 100 or mental status change (evidence of shock)

Exclusion Criteria:

Patients with any injuries above the clavicle or head injuries will be excluded. If known at the time of randomization the investigator will exclude all known minors under the age of 18, known pregnant women, and known prisoners. Patients with isolated blunt mechanism of injury such as motor vehicle accidents will be excluded. However, patients with combined blunt and penetrating torso injury will be included.

1. Injury above the clavicle
2. Isolated injury distal to the elbows or knees
3. Known age <18, pregnant, or prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival to hospital discharge | 48 hours
  Mortality at 48 hours

SECONDARY OUTCOMES:
Transfusion requirement | 48 hours
  Absence or presence of needing a transfusion
Ventilator days | 48 hours
  Absence or presence of needing a ventilator
Hospital & ICU length of stay | 48 hours
  Total time spent in hospital & ICU
Cost of hospital admission | 48 hours
  Total cost of admission
Discharge disability | 48 hours
  Absence or presence of disability

CONTACTS AND LOCATIONS:
Overall Officials: Amy Goldberg, MD, Principal Investigator — Temple University Hospital
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No